CLINICAL TRIAL: NCT03329404
Title: Evaluate the Efficacy and Safety of RBCs Derived From Mirasol-treated Whole Blood Compared With Conventional RBCs in Patients Requiring Chronic Transfusion Support
Brief Title: Efficacy and Safety of RBCs Derived From Mirasol-treated Whole Blood in Patients Requiring Chronic Transfusion (PRAISE)
Acronym: PRAISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to blood supply challenges. Subsequently approved by FDA to reopen but will not do so because of changing clinical need.
Sponsor: Terumo BCTbio (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Joint Warfighter Medical Research Program (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTS-5056
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Transfusion Dependent Thalassemia
Keywords: Thalassemia; pathogen reduction therapy
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Mirasol Red Blood Cells (MIR RBCs) (Experimental): MIR RBCs: RBCs will be derived from WB collected in CPD solution, treated with the Mirasol System for WB, LR, and stored in AS-3 for ≤ 21 days at 1-6°C
  Interventions: Device: Mirasol Red Blood Cells (MIR RBCs)
- Reference Red Blood Cells (REF RBCs) (Active Comparator): Reference Red Blood Cells (REF RBCs); LR apheresis RBCs or WB-derived RBCs will be per site standard inventory
  Interventions: Device: Reference Red Blood Cells (REF RBCs)

INTERVENTIONS:
Device: Mirasol Red Blood Cells (MIR RBCs) — Mirasol Red Blood Cells (MIR RBCs) derived from Mirasol-treated WB; WB will be Mirasol treated, centfifuged and leukoreduced and the derived RBCs will be stored before transfusion for up to 21 days and transfused according to the patient's transfusion schedule.
  Arms: Mirasol Red Blood Cells (MIR RBCs)
Device: Reference Red Blood Cells (REF RBCs) — Reference Red Blood Cells (REF RBCs) will be acquired from routine use inventory and transfused according to the patient's transfusion schedule.
  Arms: Reference Red Blood Cells (REF RBCs)

SUMMARY:
This is a prospective, multi-center, randomized, crossover trial to evaluate the clinical effectiveness of red blood cells (RBCs) derived from Mirasol-treated whole blood (WB) versus conventional RBCs in transfusion dependent thalassemia patients. Throughout the clinical study, RBC transfusion volume and frequency will be determined by each subject's treating physician.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive either Mirasol-treated RBCs followed by conventional RBCs, or to receive conventional RBCs followed by Mirasol-treated RBCs. The blood centers will collect the donor RBCs and supply the Mirasol-treated RBCs to the hospital sites for transfusion into patients. Hospital sites will order conventional RBCs as per their normal process, from their standard vendor.

Blood transfusion is the mainstay of care for individuals with thalassemia major. The purpose of transfusion is twofold: to improve the anemia and to suppress the ineffective erythropoiesis. A transfusion episode for these thalassemia patients are the routine transfusions administered on a regular schedule for the life of the patient.

The crossover trial design will consist of 2 treatment periods: Period 1 = Mirasol-treated RBCs followed by conventional (reference) RBCs; Period 2 = Reference RBCs followed by Mirasol-treated RBCs. Each period will include a 50 day wash-in phase (Day 0 of the wash-in = Day 0 of the treatment period) followed by 2 transfusion episodes. An end of study treatment follow-up visit will occur 2-4 weeks after the last per protocol transfusion, prior to the next standard of care transfusion. A final study visit will occur at least 60 days after the last per protocol transfusion.

The primary objective of the PRAISE study is to determine if percent survival of RBCs derived from Mirasol-treated WB is non-inferior to conventional RBCs when transfused into patients requiring chronic RBC transfusion support. The secondary objectives include comparing other efficacy and safety endpoints between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Transfusion dependent thalassemia patient with mean 2-4 week transfusion intervals for the prior 6 months.

  2. Age ≥ 12 years.

  3. Negative pregnancy test for women of childbearing potential and agreement to practice a medically acceptable contraception regimen throughout the participation in the clinical trial. Not required if female subjects are not of child-bearing potential (ie, prior to menses onset, surgically sterilized, 1-year postmenopausal).

  4. Signed informed consent from the patient, or if the patient is < 18 years of age, signed assent from patient and consent from parent/guardian, according to local Institutional Review Board/Ethics Committee (IRB/EC) requirements.

Exclusion Criteria:

1. Historical RBC transfusion requirement of more than 250 mL/kg/year.
2. Presence of RBC antibodies that make procurement of compatible RBC units not feasible per the treating physician's clinical judgment for reasonable execution of the study.
3. Prior treatment with pathogen-reduced RBCs with subsequent development of known antibodies to the associated RBCs.
4. Planned treatment requirement of frozen RBC products.
5. Treatment requirements for any medication that is known to cause hemolysis.
6. Receiving cardiac medications for heart failure.
7. Patients anticipated to receive massive transfusion, per the treating physician's clinical judgment.
8. Known HIV infection (defined as HIV RNA positive) with changes to antiviral regimen within the 12 months prior to screening.
9. Acute or chronic medical disorder that, in the opinion of the Investigator, would impair the ability of the patient to receive study treatment.
10. Participation in another clinical study, either concurrently or within the previous 28 days, in which the study drug or device may influence study endpoints or patient safety, according to Investigator discretion.
11. Participation in another clinical study within the past 3 months if investigational RBCs or treatment or drugs were received that are likely to have long term effect on RBCs function.
12. Pregnant or breastfeeding.
13. Planned concurrent treatment with other pathogen reduction treated blood products during participation in this study.
14. Patients who received prior treatment with pathogen-reduced RBCs within the past 120 days.
15. Inability to comply with study procedures and/or follow-up.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Cosgriff, MD, Study Director — Terumo BCT; Steve Sloan, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (9):
- United States (4):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Weill-Cornell Medical College, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Hadassah Ein Kerem Hospital, Jerusalem
- Italy (2):
  - Centro della Microcitemia ed Anemie Congenite Ospedale Gallieria, Genova, Genoa
  - U.O.C. di Ematologia e Malattie Rare del Sangue e degli Organi Ematopoietici V. Cervello Hospital, Palermo
- Ege University Children's Hospital, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine subjects were enrolled and assigned into treatment arms. The first subject signed consent on 12 April 2018 and the last subject signed consent on 03 October 2018.
Pre-assignment Details: This was a crossover study, all 9 randomized subjects were to receive both Mirasol and Reference RBCs in either period 1 or 2. 4 subjects were randomized to the MIR/REF RBC treatment sequence and 5 subjects were randomized to the REF/MIR RBC sequence. 4 subjects completed period 1, no subjects completed period 2 due to study suspension. Because no subjects completed the study, the primary endpoint was not evaluated and results are summarized by treatment type rather than treatment sequence.
Groups:
- Mirasol Red Blood Cells (MIR RBCs) Followed by Reference RBCs (REF RBCs): MIR RBCs: RBCs were derived from whole blood (WB) collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, Leukoreduced (LR), and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
  REF RBCs: LR apheresis RBCs or WB-derived RBCs were per site standard inventory.
- Reference Red Blood Cells (REF RBCs) Followed by Mirasol RBCs (MIR RBCs): REF RBCs: Leukoreduced (LR) apheresis RBCs or whole blood (WB)-derived RBCs were per site standard inventory.
  MIR RBCs: RBCs were derived from WB collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, LR, and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
Period: Overall Study
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) Followed by Reference RBCs (REF RBCs) | Reference Red Blood Cells (REF RBCs) Followed by Mirasol RBCs (MIR RBCs)
Started | 4 | 5
Completed (4 subjects were randomized to the MIR/REF RBC treatment sequence, 3 of the 4 subjects completed the first arm of the study and 1 subject did not complete the first arm of the study. 5 subjects were randomized to the REF/MIR RBC treatment sequence, 1 of the 5 subjects completed the first arm of the study and 4 subjects did not complete the first arm of the study. In summary- no subjects completed the entire study and 4 subjects completed one arm of the study.) | 3 | 1
Not Completed | 1 | 4
Not completed — The study was suspended. | 1 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized subjects.
Groups:
- Mirasol Red Blood Cells (MIR RBCs)/Reference Red Blood Cells (REF RBCs) Treatment Sequence: MIR RBCs: RBCs were derived from whole blood (WB) collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, Leukoreduced (LR), and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
  REF RBCs: LR apheresis RBCs or WB-derived RBCs were per site standard inventory.
- Reference Red Blood Cells (REF RBCs)/Mirasol Red Blood Cells (MIR RBCs) Treatment Sequence: REF RBCs: Leukoreduced (LR) apheresis RBCs or whole blood (WB)-derived RBCs were per site standard inventory.
  MIR RBCs: RBCs were derived from WB collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, LR, and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
- Total: Total of all reporting groups
Arm/Group | Mirasol Red Blood Cells (MIR RBCs)/Reference Red Blood Cells (REF RBCs) Treatment Sequence | Reference Red Blood Cells (REF RBCs)/Mirasol Red Blood Cells (MIR RBCs) Treatment Sequence | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Normalized Hemoglobin (Hb AUC) Calculated From Normalized Hb Between Successive Transfusions as a Measure of Percent Surviving RBCs
Description: The Hb AUC is calculated using the trapezoidal method on normalized Hb. The normalization is accomplished by dividing all posttransfusion Hb values by the 15-minute posttransfusion Hb level. The ratio is expressed as a percentage. A natural log-transform of the observed normalized Hb AUC will be utilized.
Time Frame: Crossover design with 2 treatment periods. Each period included a 50-day wash-in followed by 2 transfusion episodes for primary endpoint assessment. Expected participation was approximately 7-10 months, depending on the subject's transfusion schedule.
Population: The Statistical Analysis Plan was not executed for this study because the study was stopped prematurely. Ninety-seven subjects were planned to be enrolled however 9 were randomized. None of the 9 randomized subjects completed the sequence arms and met the per protocol criteria and as such the primary endpoint was not collected.
Groups:
- Mirasol Red Blood Cells (MIR RBCs): MIR RBCs: RBCs were derived from whole blood (WB) collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, Leukoreduced (LR), and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
  REF RBCs: LR apheresis RBCs or WB-derived RBCs were per site standard inventory.
- Reference Red Blood Cells (REF RBCs): REF RBCs: Leukoreduced (LR) apheresis RBCs or whole blood (WB)-derived RBCs will be per site standard inventory.
  MIR RBCs: RBCs will be derived from WB collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, LR, and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hb Increment
Description: (post-transfusion Hb - pre-transfusion Hb)/Hb transfused]/RBC volume in subject at pre-transfusion
Time Frame: Endpoint assessments was evaluated at 15 min Post Transfusion, 1 Day Post Transfusion, 7 Day Post Transfusion, and End of Transfusion Episode.
Population: The Statistical Analysis Plan was not executed for this study because the study was stopped prematurely. Ninety-seven subjects were planned to be enrolled however 9 were randomized. None of the 9 randomized subjects completed the sequence arms and met the per protocol criteria and as such the secondary endpoint was not analyzed as planned in the Statistical Analysis Plan.
  The limited data collected was analyzed per intervention, not by sequence.
Measure: Mean (Standard Deviation); unit: delta g/dl per mL RBC transfused
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 4 | 8
delta g/dl per mL RBC transfused
  15 minute Post-Transfusion | 0.000299 (0.000422) | 0.000288 (0.000400)
  1 Day Post-Transfusion | 0.000297 (0.000486) | 0.000362 (0.000330)
  7 Day Post-Transfusion | 0.000173 (0.000287) | 0.000149 (0.000181)
  End of Transfusion Interval | 0.000014 (0.000159) | -0.000041 (0.0000999)

3. Secondary Outcome: Actual Hb Level Post-transfusion (15 Min)
Description: Actual Hb level post-transfusion (15 min)
Time Frame: An average of 30 weeks consisting of 2 crossover treatment periods with each period including a 50 day wash-in phase followed by 2 transfusion episodes for endpoint assessment
Population: The SAP was not executed for this study as the study was stopped prematurely. None of the 9 randomized subjects completed the sequence arms and met the per protocol criteria. Post-hoc analysis was performed by intervention, not by the randomized sequence arm. Of the 9 randomized subjects, 1 subject did not enter either treatment period.There were 4 MIR treatment periods and 8 REF treatment periods.
Measure: Mean (Standard Deviation); unit: grams/dL
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 4 | 8
grams/dL | 11.19 (1.44) | 11.49 (0.65)

4. Other Pre Specified Outcome: Percentage Decline in Post-transfusion Hb Level
Description: Percentage decline in post-transfusion Hb level
Time Frame: as for outcome 3
Population: The Statistical Analysis Plan was not executed for this study because the study was stopped prematurely. Ninety-seven subjects were planned to be enrolled however 9 were randomized. None of the 9 randomized subjects completed the sequence arms and met the per protocol criteria and as such the secondary endpoint was not analyzed according to the Statistical Analysis Plan. The limited data collected was analyzed per intervention, not by sequence.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 4 | 8
percent change | -4.256 (5.367) | -3.249 (5.568)

5. Other Pre Specified Outcome: RBC Mass Infused
Description: volume x Hb/unit
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 4 | 8
grams | 1445.796 (33.622) | 107.039 (29.583)

6. Other Pre Specified Outcome: Number of Antibody Screening Test With Confirmed Specificity to RBCs Derived From Mirasol-treated WB
Description: Antibody screening was performed in a total of 8 (100%) subjects in the SS at a total of 97 intervals (Pre-Transfusion, 7 Days Post-Transfusion or End of Study Treatment Follow-up Visit).
Time Frame: Up to 40 weeks consisting of 2 crossover treatment periods with each period including a 50 day wash-in phase followed by 2 transfusion episodes for endpoint assessment and a final study visit 60 days after last study transfusion
Population: Safety Set. The Statistical Analysis Plan was not executed for this study because the study was stopped prematurely. Of the 97 subjects planned to be enrolled, only 9 subjects were randomized and none completed the sequence arms. Of the 9 subjects, one did not enter either treatment period. The limited data collected was analyzed per intervention, not by sequence.
Measure: Count of Units; unit: antibody screen test
Units Other Than Participants: antibody screen test
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
Number analyzed (Participants) | 4 | 8
Number analyzed (antibody screen test) | 43 | 54
antibody screen test | 0 | 3

7. Other Pre Specified Outcome: Number of Participants With Human Leukocyte Antigen (HLA) Alloimmunization Post Transfusion
Description: The highest of three different normalized background ratio (NBG) cut-offs was used to quantify positivity for Class I HLA antibodies prior to transfusion as it was used to identify conversion from HLA antibody negative prior to transfusion to positivity after transfusion(s) within the applicable treatment group.
Time Frame: Up to 40 weeks consisting of 2 crossover treatment periods with each period including a 50 day wash-in phase followed by 2 transfusion episodes for endpoint assessment and a final study visit 60 days after last study.
Population: Safety Set. The Statistical Analysis Plan was not executed for this study because the study was stopped prematurely. Of the 97 subjects planned to be enrolled, only 9 subjects were randomized and none completed the sequence arms. Of the 9 subjects, one did not enter either treatment period. The limited data collected was analyzed by sequence.
Measure: Count of Participants; unit: Participants
Groups:
- Mirasol Red Blood Cells (MIR RBCs)/ Reference RBCs (REF RBCs) Treatment Sequence: MIR RBCs: RBCs were derived from whole blood (WB) collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, Leukoreduced (LR), and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
  REF RBCs: LR apheresis RBCs or WB-derived RBCs were per site standard inventory.
- Reference Red Blood Cells (REF RBCs)/Mirasol RBCs (MIR RBCs) Treatment Sequence: REF RBCs: Leukoreduced (LR) apheresis RBCs or whole blood (WB)-derived RBCs will be per site standard inventory.
  MIR RBCs: RBCs will be derived from WB collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, LR, and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
Arm/Group | Mirasol Red Blood Cells (MIR RBCs)/ Reference RBCs (REF RBCs) Treatment Sequence | Reference Red Blood Cells (REF RBCs)/Mirasol RBCs (MIR RBCs) Treatment Sequence
Number analyzed (Participants) | 4 | 4
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: This was a crossover study, therefore adverse events are reported by treatment received, some subjects received both treatments. Of the 9 randomized subjects, 1 subject did not receive any study transfusions, 4 of the 9 subjects received some MIR RBC transfusions and 8 of the 9 subjects received some REF RBC transfusions.
Groups:
- Mirasol Red Blood Cells (MIR RBCs): MIR RBCs: RBCs were derived from whole blood (WB) collected in citrate phosphate dextrose (CPD) solution, treated with the Mirasol System for WB, leukoreduced, and stored in Additive Solution Formula 3 (AS-3) for ≤ 21 days at 1 - 6°C.
- Reference Red Blood Cells (REF RBCs): REF RBCs: Leukoreduced apheresis RBCs or whole blood-derived RBCs were per site standard inventory.
Arm/Group | Mirasol Red Blood Cells (MIR RBCs) | Reference Red Blood Cells (REF RBCs)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 1/4 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirasol Red Blood Cells (MIR RBCs) (N=4) | Reference Red Blood Cells (REF RBCs) (N=8)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary endpoint was not evaluated due to the early termination of the study and subsequent small sample size with no subjects completing both Period 1 and Period 2 of the study preventing any meaningful results. Due to the limited dataset we were not able to make any meaningful inferences and as such the data should be viewed with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03329404/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03329404/SAP_001.pdf